CLINICAL TRIAL: NCT01142700
Title: A Randomized, Placebo-controlled, Phase 2a Study of BMS-824393 in Combination With Peginterferon Alfa-2a (Pegasys) and Ribavirin (Copegus) in Treatment Naive Subjects With Chronic Hepatitis C Virus Genotype I
Brief Title: A Study of BMS-824393 in Combination With Peginterferon Alfa-2a (Pegasys) and Ribavirin (Copegus) in Treatment Naive Subjects With Chronic Hepatitis C Virus Genotype I
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AI451-004; 2010-018702-36 (EudraCT Number)
Record Dates: First submitted 2010-06-03; First posted 2010-06-11 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Hepatitis C Virus Genotype 1
MeSH Terms: interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- BMS-824393 (10mg) (Experimental): Plus Peginterferon Alfa-2a and Ribavirin
  Day 1 - Week 12
  Interventions: Drug: BMS-824393; Drug: Peginterferon Alpha-2a; Drug: Ribavirin
- BMS-824393 (30 mg) (Experimental): Plus Peginterferon Alfa-2a and Ribavirin
  Day 1 - Week 12
  Interventions: Drug: BMS-824393; Drug: Peginterferon Alpha-2a; Drug: Ribavirin
- BMS-824393 (100 mg) (Experimental): Plus Peginterferon Alfa-2a and Ribavirin
  Day 1 - Week 12
  Interventions: Drug: BMS-824393; Drug: Peginterferon Alpha-2a; Drug: Ribavirin
- Placebo (Placebo Comparator): Plus Peginterferon Alfa-2a and Ribavirin
  Day 1 - Week 12
  Interventions: Drug: Placebo; Drug: Peginterferon Alpha-2a; Drug: Ribavirin
- Peginterferon alfa-2a plus Ribavirin (Other): Weeks 13 - 48
  Interventions: Drug: Peginterferon Alpha-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: BMS-824393 — Capsule, Oral, 10 mg, once daily
  Arms: BMS-824393 (10mg)
Drug: BMS-824393 — Capsule, Oral, 30 mg, once daily
  Arms: BMS-824393 (30 mg)
Drug: BMS-824393 — Capsule, Oral, 100 mg, once daily
  Arms: BMS-824393 (100 mg)
Drug: Placebo — Capsule, Oral, 0 mg, once daily
  Arms: Placebo
Drug: Peginterferon Alpha-2a — Syringe, subcutaneous 180 mcg/0.5 mL, weekly
  Other Names: Pegasys
Drug: Ribavirin — Tablet, Oral, 400 or 600 mg based on weight (am) and 600 mg (pm), twice daily
  Other Names: Copegus

SUMMARY:
Based on 12-week on-treatment data, at least 1 dose of BMS-824393 can be identified which is safe, well tolerated, and has sufficient antiviral activity to progress to late stage clinical trials when combined with pegIFNα/RBV for treatment of chronically infected hepatitis C virus genotype 1 treatment-naive subjects.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive subjects with genotype 1 chronic HCV
* HCV RNA ≥ 100,000 IU/mL at screening
* Seronegative for HIV and HBsAg
* Liver biopsy within prior 2 years demonstrating no cirrhosis

Exclusion Criteria:

* Any evidence of liver disease other than hepatitis C
* Diagnosed or suspected hepatocellular carcinoma
* Laboratory values: neutrophil count < 1500 cells/μL, platelet count < 90,000/μL; Hemoglobin ≤ 12 g/dL (120g/L) for women and ≤ 13 g/dL (130 g/L) for men
* Cirrhosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by the frequency of serious adverse events (SAEs) and discontinuations due to adverse events (AEs) | Week 4
Safety as measured by the frequency of serious adverse events (SAEs) and discontinuations due to adverse events (AEs) | Week 12
Safety as measured by the frequency of serious adverse events (SAEs) and discontinuations due to adverse events (AEs) | Week 24
Safety as measured by the frequency of serious adverse events (SAEs) and discontinuations due to adverse events (AEs) | Week 48
Antiviral activity as determined by the proportion of subjects with extended rapid virologic response (eRVR) defined as undetectable HCV RNA | Week 4
Antiviral activity as determined by the proportion of subjects with extended rapid virologic response (eRVR) defined as undetectable HCV RNA | Week 12

SECONDARY OUTCOMES:
Proportion of subjects with rapid virologic response (RVR), defined as undetectable RNA | Week 4
Proportion of subjects with complete early virologic response (cEVR), defined as undetectable HCV RNA | Week 12
Proportion of subjects with a sustained virologic response (SVR), defined as HCV RNA undetectable | Week 12 (SVR12)
Proportion of subjects with a sustained virologic response (SVR), defined as HCV RNA undetectable | Week 24 (SVR24)
Resistant variants associated with virologic failure | Week 4
Resistant variants associated with virologic failure | Week 12
Resistant variants associated with virologic failure | Follow up Week 12
Resistant variants associated with virologic failure | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (11):
- United States (11):
  - Local Institution, Coronado, California
  - Research And Education, Inc., San Diego, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Bach And Godofsky Infectious Diseases, Bradenton, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Vita Medical Center & Research Solutions, Inc., Tamarac, Florida
  - Gastrointestinal Specialists Of Georgia Pc, Mareitta, Georgia
  - Maryland Digestive Disease Research, Laurel, Maryland
  - Local Institution, Philadelphia, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - Liver Institute Of Virginia Bon Secours Health System, Newport News, Virginia

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx